CLINICAL TRIAL: NCT07087769
Title: Optimizing Post-Stroke Gait Symmetry: Integrating Mechanical Constraints and Sensory Feedback to Enhance Paretic Leg Propulsion
Brief Title: Optimizing Gait Symmetry After Stroke Using Mechanical Constraints and Sensory Feedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25-0102
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Split-belt Treadmill; Resistance Exercise; Feedback; Gait Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will undergo multiple gait training conditions in a single session, including combinations of treadmill walking (tied-belt and split-belt), backward resistance (pelvis, ankle, or both), and sensory feedback (visual, auditory, or combined). All participants will receive all conditions in a within-subject crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait Training with Combined Sensory Feedback and Mechanical Constraints (Experimental): All participants will receive various gait training conditions during a single session. Conditions include treadmill walking (tied-belt and split-belt), backward-directed resistance (applied at pelvis, ankle, or both), sensory feedback (visual, auditory, or combined), and a final combined condition integrating both resistance and feedback. This is a within-subject crossover design.
  Interventions: Behavioral: Treadmill Walking with Split-Belt and/or Tied-Belt Conditions; Behavioral: Mechanical Resistance (Pelvis and/or Ankle) depending on participant's walking capacity; Behavioral: Sensory Feedback Training

INTERVENTIONS:
Behavioral: Treadmill Walking with Split-Belt and/or Tied-Belt Conditions — Participants will walk on an instrumented treadmill under split-belt and/or tied-belt conditions depending on their walking capacity. The belt speeds will be adjusted to facilitate locomotor adaptation and evaluate propulsion symmetry.
Behavioral: Mechanical Resistance (Pelvis and/or Ankle) depending on participant's walking capacity — Participants will walk on a treadmill (Split-belt and/or Tied-belt) with backward-directed resistance applied at the pelvis, ankle, or both. The resistance is used to challenge paretic leg propulsion and assess adaptive gait responses.
Behavioral: Sensory Feedback Training — Real-time feedback-visual, auditory, or combined-will be provided based on the propulsive force generated during split-belt and/or tied-belt treadmill walking, with or without mechanical resistance.

SUMMARY:
This single-session study aims to evaluate a novel gait training protocol that integrates mechanical constraints and sensory feedback to enhance paretic leg propulsion in individuals post-stroke. The study will include 15 individuals who have experienced a stroke and 15 healthy adults, each aged 20 years or older. Participants will walk on both tied-belt and split-belt treadmills under various training conditions, including backward-directed resistance (applied at the pelvis, ankle, or both) and real-time sensory feedback (visual, auditory, or combined). These interventions will be applied individually and in combination to identify the most effective environment for promoting symmetrical gait patterns. Each session will last approximately two hours. The equipment used is non-invasive, and the risk to participants is minimal.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of an integrated gait training paradigm that combines mechanical task constraints and sensory feedback during split-belt treadmill walking to enhance paretic leg propulsion and improve propulsion symmetry in individuals post-stroke. The risks associated with this study are lower than those encountered during daily walking in the community and in typical physical therapy clinics, where patients with physical impairments routinely engage in challenging exercises to improve their abilities. There is a slight possibility of local skin irritation or rash resulting from the non-allergenic adhesive tape or sensor gel used to attach the EMG sensors. This is a rare occurrence and typically resolves within one to two days without medical intervention.

This study will last approximately one to two hours, depending on your condition, and involves a one-time visit.

If you choose to participate in this study, the participant will be asked to:

1. Sign a consent form approved by the University of Texas Medical Branch IRB, outlining the study's purpose, procedures, benefits, risks, and policies.
2. Share medical history and well-being, and have weight, height, and heart rate (via smartwatch) monitored.
3. Assess your walking capacity.
4. Assess the Optimal Gait Training Protocol using Treadmill, Sensory Feedback, and Mechanical task constraints.

ELIGIBILITY:
Inclusion Criteria:

Aged 20 years or older

For stroke group: clinical diagnosis of stroke at least 1 month prior to participation

Ability to walk at least 10 meters with or without assistive devices

For healthy group: able to walk independently without assistive devices

Exclusion Criteria:

Life expectancy less than one year

Comatose or unable to follow three-step commands

Amputation of any lower limb

Poorly controlled diabetes (e.g., foot ulceration)

Blindness

Progressive neurological disease

Medically unstable condition

Significant musculoskeletal impairments affecting gait

Congestive heart failure or unstable angina

Peripheral vascular disease

Severe neuropsychiatric conditions (e.g., dementia, cognitive deficits, severe depression)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Paretic Leg Propulsive Force | Within a single session (approximately 2 hours)
  Peak anterior ground reaction force of the paretic leg will be measured using an instrumented split-belt treadmill . Changes in propulsive force under different treadmill and resistance/feedback conditions will be analyzed to evaluate improvements in gait symmetry.

SECONDARY OUTCOMES:
Muscle Activity of Lower Extremity During Treadmill and overgrouun Walking | Day 1 (during treadmill and overground walking trials)
  Surface EMG (Delsys Inc.) will be used to measure activity of major lower limb muscles (e.g., Tibialis anterior and soleus) during treadmill walking under different resistance and feedback conditions.
Step Length (m) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Step length (in meters) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average step length for each participant will be reported.
Hip Joint Range of Motion (degrees) During Treadmill Walking Using Vicon Motion Capture System | Day 1 (during treadmill walking trials)
  Hip joint range of motion (ROM), measured in degrees, will be assessed using the Vicon motion capture system during treadmill walking on Day 1. ROM will be defined as the difference between peak flexion and peak extension angles in the sagittal plane. Kinematic data will be collected across multiple gait cycles, and the average ROM per participant will be reported.
Walking Speed (m/s) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Walking speed (in meters per second) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average walking speed for each participant will be reported.
Cadence (steps/min) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Cadence (in steps per minute) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average cadence will be reported per participant.
Swing Time (s) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Swing time (in seconds) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average swing time per leg will be reported per participant.
Stance Time (s) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Stance time (in seconds) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average stance time per leg will be reported per participant.
Stride Length (m) During Overground Walking Using Zeno Walkway | Day 1 (during overground walking trials)
  Stride length (in meters) will be measured using the Zeno Walkway Gait Analysis System during overground walking trials on Day 1. The average stride length per participant will be reported.
Knee Joint Range of Motion (degrees) During Treadmill Walking Using Vicon Motion Capture System | Day 1 (during treadmill walking trials)
  Knee joint range of motion (ROM), measured in degrees, will be assessed using the Vicon motion capture system during treadmill walking on Day 1. ROM will be defined as the difference between peak flexion and peak extension angles in the sagittal plane. Multiple gait cycles will be analyzed, and the average ROM per participant will be reported.
Ankle Joint Range of Motion (degrees) During Treadmill Walking Using Vicon Motion Capture System | Day 1 (during treadmill walking trials)
  Ankle joint range of motion (ROM), measured in degrees, will be assessed using the Vicon motion capture system during treadmill walking on Day 1. ROM will be calculated as the difference between peak dorsiflexion and peak plantarflexion angles in the sagittal plane. Data from multiple gait cycles will be averaged and reported per participant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No